CLINICAL TRIAL: NCT00433225
Title: Efficacy of Topical Ketorolac Versus Placebo for Improving Visual Outcomes Following Multifocal IOL Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5293
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Macula Thickening
MeSH Terms: interventions — prednisolone acetate

INTERVENTIONS:
Drug: Prednisolone Acetate
Drug: Ketorolac 0.4%
Drug: Gatifloxacin 0.3%

SUMMARY:
The purpose of this study was to evaluate the efficacy of ketorolac 0.4% on quality of vision and macula thickening in patients undergoing cataract surgery using the ReStor® multifocal IOL.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 50 years old
* Scheduled to undergo bilateral phacoemulsification with implantation of a multifocal IOL.
* Likely to complete all study visits and able to provide informed consent
* Visual potential of 20/25 or better

Exclusion Criteria:

* · Prior use of topical ketorolac

  * Known contraindications to any study medication or ingredients
  * Active ocular diseases or uncontrolled systemic disease
  * Active ocular allergies

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of Long Island, Rockville Centre, New York, United States